CLINICAL TRIAL: NCT00862602
Title: Type 2 Diabetes Risk in Women With Gestational Diabetes
Brief Title: Pedometers for Gestational Diabetes
Acronym: PEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Catherine Kim, associate professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23DK071552 (NIH); K23DK071552 (NIH); R03DK083332 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes
Keywords: GDM; gestational diabetes; pregnancy; diabetes; walking; exercise; pedometer; online
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stepping Up to Health
  Interventions: Behavioral: Stepping Up to Health
- 2 (No Intervention): Usual care group

INTERVENTIONS:
Behavioral: Stepping Up to Health — Internet-mediated pedometer-based intervention with gradually increasing goals and feedback on step counts. Also includes educational content targeted at women who have had gestational diabetes about exercise, diet & nutrition and prevention.
  Arms: 1

SUMMARY:
Ten to 50% of women with gestational diabetes (GDM), or glucose intolerance first recognized during pregnancy, develop diabetes within 5 years after delivery. Although intensive interventions can reduce diabetes incidence in women with impaired glucose tolerance, it is unknown if such strategies would be effective in women with GDM. Women with recent GDM, even though no longer pregnant, face significant barriers to lifestyle modification, including caregiving responsibilities and low perception of risk. Web-based programs can reinforce physical activity through visual feedback of pedometer output, tailored messaging, education, and on-line communities. Such a program is currently available for adults with chronic disease and is led by Dr. Richardson, a co-PI on this application. Using data from focus group and survey work conducted by Dr. Kim, the other co-PI, this program can be modified to women with recent GDM. For Specific Aim 1, we propose to adapt a chronic disease web-based pedometer program to women with recent GDM. For Specific Aim 2, we propose to conduct a pilot and feasibility study of the program. The intervention will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes diagnosis within past three years
* Access to computer with internet, USB port and Windows XP or Vista
* Regular email user (weekly or more)
* Can walk a block on her own
* Sedentary (less than 150 minutes purposeful physical activity per week)

Exclusion Criteria:

* Pregnancy
* Unable to consent legally

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Weight loss | Pre-post
Glucose tolerance | Pre-Post

SECONDARY OUTCOMES:
Hemoglobin A1c | Pre-post
Step counts | Pre-Post
Insulin | Pre-post

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Kim, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States